CLINICAL TRIAL: NCT00695994
Title: The Effect of Pharmacogenetics on Treatment Toxicities and Outcomes in East Asian and Caucasian Patients Undergoing Docetaxel or Gemcitabine-based Chemotherapy
Brief Title: The Effect of Docetaxel or Gemcitabine-based Chemotherapy in East Asian and Caucasian Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Ross Soo, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRG-PG02/26/06
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Non Small Cell Lung Cancer; Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — Docetaxel; Gemcitabine; Carboplatin

ARMS (2):
- Docetaxel (Experimental): Docetaxel will be administered at a dose of 75 mg/m2 given as a 1-hour intravenous infusion on day 1 of a 21-day cycle.
  Interventions: Drug: Docetaxel
- Gemcitabine and carboplatin (Experimental): Carboplatin will be administered as a 1-hour infusion on day 1 of a 21-day cycle. Gemcitabine will be administered as a 30-minute infusion at the dose of 1000 mg/m2 in 250 mL over 30 minutes, on day 1 and 8 of a 21-day cycle. It will be given after carboplatin infusion.
  Interventions: Drug: gemcitabine and carboplatin

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be administered at a dose of 75 mg/m2 given as a 1-hour intravenous infusion on day 1 of a 21-day cycle. Docetaxel is re-constituted in 500 mL of normal saline and infused through a peripheral or central venous line. Docetaxel (Taxotere®, Sanofi-Aventis Inc.) is available in 80 mg and 20 mg in 2 mL polysorbate 80, 13% (w/w) ethanol in Water for Injection.
  Other Names: Docetaxel (Taxotere®, Sanofi-Aventis Inc.)
  Arms: Docetaxel
Drug: gemcitabine and carboplatin — Gemcitabine (Gemzar®, Lily Inc.) is available in vials containing 1000 mg or 200 mg of active drug formulated with mannitol (200 mg or 1 g, respectively) and sodium acetate (12.5 mg or 62.5 mg, respectively) as a sterile lyophilized powder.
  Carboplatin (Spectrum Pharmaceuticals, Inc.) is supplied as a 10 mg/mL aqueous solution. Unopened vials of gemcitabine are stable when stored at controlled room temperature at 25°C, protected from bright light. It can be diluted in normal saline or 5% dextrose. The solution remains stable for 8 hours at 25°C after reconstitution.
  Carboplatin will be administered as a 1-hour infusion on day 1 of a 21-day cycle. It will be given before gemcitabine at the dose to achieve an AUC of 5 using the Calvert formula.
  Gemcitabine will be administered as a 30-minute infusion at the dose of 1000 mg/m2 in 250 mL over 30 minutes, on day 1 and 8 of a 21-day cycle. It will be given after carboplatin infusion.
  Other Names: Gemcitabine (Gemzar®, Lily Inc.); Carboplatin (Spectrum Pharmaceuticals, Inc.)
  Arms: Gemcitabine and carboplatin

SUMMARY:
The aims of this study are:

1. to compare the toxicity profile and efficacy of gemcitabine/carboplatin or docetaxel in East Asian and Caucasian patients.
2. to determine the genotype distribution of genes involved in docetaxel and gemcitabine pathways in East Asian and Caucasian patients.
3. to evaluate the association between genotypes and

   1. treatment toxicity
   2. treatment efficacy
   3. pharmacokinetics.

DETAILED DESCRIPTION:
Germline polymorphisms are inherited genetic variations present in all cells of the body. Mounting evidence has shown that genetic polymorphisms in drug metabolizing, transporter and targets genes are major determinants of response to drugs.

The aims of this study are to compare (i) the toxicity profile and efficacy of gemcitabine/carboplatin or docetaxel, (ii) the distribution of genes involved in docetaxel and gemcitabine pathways and (iii) to evaluate the association between pharmacogenetics, pharmacokinetics and pharmacodynamics in East Asian and Caucasian patients.

To date, most pharmacogenetic strategies are predominantly focused on the role of single genes, in the regulation of drug metabolism. However, there is clear evidence that treatment outcomes are under the control of a network of genes, each contributing to the patient's phenotype. In this study, we propose taking a global approach to include relevant candidate genes in drug pathways to evaluate the effect of polymorphisms and treatment outcomes. We have selected two commonly used chemotherapy regimens based on our previous observation of interethnic variability in treatment outcomes and candidate polymorphisms.

By incorporating pharmacokinetic (drug level, drug elimination etc), pharmacodynamic (treatment response, survival etc) and pharmacogenetic approaches in clinical trials, it would enhance our understanding of the inter-individual variability in response and toxicity to drug treatment, and is the first step towards individualized drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed i) AJCC/UICC stage IIIB or IV non small cell lung cancer and stage IV breast cancer for which docetaxel is indicated. ii) AJCC/UICC stage IIIB or stage IV non small cell lung cancer for which gemcitabine/carboplatin is indicated.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >=20 mm with conventional techniques or as >=10 mm with spiral CT scan. See section 11.2 for the evaluation of measurable disease.
* Eligible patients must not have been on previous anticancer therapy including chemotherapy, radiotherapy, biological therapy, or investigational therapy for at least 4 weeks before study entry (6 weeks if prior therapy included nitrosoureas or mitomycin C). Prior neoadjuvant or adjuvant chemotherapy, or chemotherapy given concurrently with radiotherapy for non- metastatic disease, is allowed if the last dose last dose was given 6 months or more before study entry.
* Patients eligible for docetaxel should have received at least one prior line of palliative chemotherapy. Patients eligible for gemcitabine/carboplatin should not have prior palliative therapies.
* Age >=18 years.
* Life expectancy of greater than 8 weeks.
* ECOG performance status <=2 (Karnofsky >=60%).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL
  * platelets >=100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >=60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients should not be receiving any other investigational agents.
* Patients with rapidly progressing brain metastases should be excluded from this clinical trial because of their poor prognosis. Furthermore they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel or gemcitabine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because docetaxel and gemcitabine are embryotoxic/fetotoxic with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with docetaxel or gemcitabine, breastfeeding should be discontinued if the mother is treated with docetaxel or gemcitabine. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Treatment toxicities | 36 weeks
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]

SECONDARY OUTCOMES:
objective tumour response, survival, median time to progression, and duration of response | 36 weeks
  All patients included in the study must be assessed for response to treatment. Each patient will be assigned one of the following categories: 1) complete response, 2) partial response, 3) stable disease, 4) progressive disease, 5) early death from malignant disease, 6) early death from toxicity, 7) early death because of other cause, or 9) unknown (not assessable, insufficient data).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Limviphuvadh V, Tan CS, Konishi F, Jenjaroenpun P, Xiang JS, Kremenska Y, Mu YS, Syn N, Lee SC, Soo RA, Eisenhaber F, Maurer-Stroh S, Yong WP. Discovering novel SNPs that are correlated with patient outcome in a Singaporean cancer patient cohort treated with gemcitabine-based chemotherapy. BMC Cancer. 2018 May 11;18(1):555. doi: 10.1186/s12885-018-4471-x. PMID 29751792